CLINICAL TRIAL: NCT00003981
Title: Phase I Study to Determine the Safety of E7070 in Patients With a Solid Tumor as a Single IV Infusion Weekly X 4, Repeated Every 6 Weeks
Brief Title: E7070 in Treating Patients With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-16975; EORTC-16975; EISAI-E7070-E044-103
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2012-07-11 (Estimated); Status verified 2012-07

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — N-(3-chloro-7-indolyl)-1,4-benzenedisulphonamide

INTERVENTIONS:
Drug: indisulam

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of E7070 in treating patients who have solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of E7070 when administered to adult patients with solid tumors.
* Determine the qualitative and quantitative toxic effects of this drug and study the predictability, duration, intensity, onset, reversibility and dose relationship of the toxic effects in this patient population.
* Propose a safe dose for phase II study.
* Assess the pharmacokinetics of this drug at different dose levels in this patient population.
* Determine any possible antitumor activity of this drug in this patient population.

OUTLINE: This is a dose escalation study.

Patients receive E7070 IV over 1 hour on days 1, 8, 15, and 22. Treatment continues every 6 weeks for at least 2 courses in the absence of unacceptable toxicity or disease progression.

Cohorts of 3-6 patients receive escalating doses of E7070 is escalated until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 6 patients experience dose limiting toxicity.

Patients are followed every 3 weeks.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study over 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed solid tumor that is not amenable to standard therapy
* No brain involvement or leptomeningeal disease

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9 g/dL

Hepatic:

* Bilirubin less than 1.5 mg/dL
* Liver function tests no greater than 2.5 times upper limit of normal (ULN) (no greater than 5 times ULN if liver metastases present)

Renal:

* Creatinine no greater than 1.4 mg/dL OR
* Creatinine clearance at least 60 mL/min

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No active bacterial infections (e.g., abscess or fistulae)
* No other nonmalignant disease that precludes protocol therapy
* No history of alcoholism, drug addiction, or psychotic disorders that preclude participation
* No glaucoma

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* At least 4 weeks since prior immunotherapy

Chemotherapy:

* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* No other concurrent antitumor drugs

Endocrine therapy:

* At least 4 weeks since prior anticancer hormonal therapy

Radiotherapy:

* At least 4 weeks since prior radiotherapy (6 weeks for extensive radiotherapy)
* No concurrent radiotherapy (except localized palliative radiotherapy)

Surgery:

* Not specified

Other:

* No concurrent sulfonylurea agent for diabetes or antiarrhythmic agents
* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 1998-04

CONTACTS AND LOCATIONS:
Overall Officials: Axel R. Hanauske, MD, PhD, MBA, Study Chair — University Hospital, Gasthuisberg
Locations (26):
- Austria (2):
  - Innsbruck Universitaetsklinik, Innsbruck
  - Kaiser Franz Josef Hospital, Vienna
- Belgium (4):
  - Institut Jules Bordet, Brussels
  - Ludwig Institute for Cancer Research, Brussels
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Herlev Hospital - University Hospital of Copenhagen, Copenhagen, Denmark
- France (5):
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Leon Berard, Lyon
  - CRLCC Nantes - Atlantique, Nantes-Saint Herblain
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif
- Universitaetsklinikum Essen, Essen, Germany
- Netherlands (5):
  - Vrije Universiteit Medisch Centrum, Amsterdam
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - University Medical Center Nijmegen, Nijmegen
  - Erasmus University Medical Center, Rotterdam
- Norwegian Radium Hospital, Oslo, Norway
- Switzerland (3):
  - University Hospital, Basel
  - Inselspital, Bern, Bern
  - Kantonsspital - St. Gallen, Sankt Gallen
- United Kingdom (4):
  - Newcastle General Hospital, Newcastle upon Tyne, England
  - Royal Marsden Hospital, Sutton, England
  - Ninewells Hospital and Medical School, Dundee, Scotland
  - Western General Hospital, Edinburgh, Scotland